CLINICAL TRIAL: NCT00693615
Title: Study to Evaluate the Safety and Immunogenicity of MEDI-517, a Virus-Like Particle Vaccine Against Human Papillomavirus Types 16 and 18, When Formulated With Aluminum Hydroxide, AS04, or Without Adjuvant, in Healthy Adult Female Volunteers
Brief Title: Safety and Immunogenicity Study of MEDI-517 (GSK 580299) With or Without Adjuvant in Healthy Adult Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 580299/004
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Papillomavirus
Keywords: HPV, Vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Formulation 1 of the vaccine (MEDI-517 HPV-16/18 VLP AS04 vaccine)
  Interventions: Biological: MEDI-517 HPV-16/18 VLP AS04 vaccine
- Group B (Experimental): Formulation 2 of the vaccine [with Al(OH)3]
  Interventions: Biological: MEDI-517 HPV-16/18 VLP vaccine with Al(OH)3
- Group C (Experimental): Formulation 3 of the vaccine (without adjuvant)
  Interventions: Biological: MEDI-517 HPV-16/18 VLP vaccine without adjuvant

INTERVENTIONS:
Biological: MEDI-517 HPV-16/18 VLP AS04 vaccine — IM injection
  Arms: Group A
Biological: MEDI-517 HPV-16/18 VLP vaccine with Al(OH)3 — IM injection
  Arms: Group B
Biological: MEDI-517 HPV-16/18 VLP vaccine without adjuvant — IM injection
  Other Names: MEDI-517 HPV-16/18 VLP AS04 vaccine; MEDI-517 HPV-16/18 VLP vaccine with Al(OH)3
  Arms: Group C

SUMMARY:
The goals of this study are to describe the safety, reactogenicity and immunogenicity of MEDI-517 with and without adjuvant in HPV-naïve humans. Long-term immune data is collected.

This study was originally performed by MedImmune. However, GSK is now responsible for the clinical development of the HPV vaccine.

DETAILED DESCRIPTION:
This is a Phase II, double-blind, randomized, comparative trial of three formulations of MEDI-517 given at 0, 30, and 180 days by intramuscular injection. The volunteers in this study will be healthy females 18 through 30 years of age. The study collects safety, reactogenicity and immunogenicity data of MEDI-517 with and without adjuvant. Extended follow-up will provide long-term immune response data.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 through 30 years of age (must not have reached the 31st birthday)
* Written informed consent obtained from the volunteer
* Unless previously surgically sterilized, agrees to use an effective method of birth control beginning 30 days before the first study injection and continuing through 60 days after the final study injection
* Must have a negative serum pregnancy test within 21 days of study entry and must not be breast feeding
* Healthy by medical history and physical examination
* Seronegative for HPV-16 and HPV-18 antibody by ELISA within 21 days of study entry
* Cervical specimen negative for high-risk HPV DNA using the Digene Hybrid Capture® II HPV test (high-risk types Probe B) within 21 days of study entry
* Normal Pap smear, using the Cytyc ThinPrep® Pap Test, within 21 days of study entry
* No evidence of anogenital HPV lesions or physical findings suggestive of other gynaecologic pathogens on pelvic examination within 21 days of study entry
* Agrees to no other vaccines or experimental therapy until 30 days after the last study injection

Exclusion Criteria:

* Acute illness or fever (oral temperature ≥ 99.5°F [37.5°C]) at start of the study
* History or clinical manifestations of significant medical or psychiatric disorder
* Use of immunosuppressive medication (inhaled and topical corticosteroids are permitted) within the previous 90 days or history of immunodeficiency
* History of cancer
* History of alcohol or drug abuse within the past 2 years
* Abnormal laboratory blood values at screening. Other abnormal laboratory values in the screening panel which in the opinion of the principal investigator are judged to be clinically significant
* Receipt of immunoglobulin or blood products within 90 days prior to study entry
* History of abnormal Pap smear (other than a single prior report of ASCUS or indeterminate Pap smear with a subsequent normal report)
* Genital herpes disease involving the cervix or with disease characterized on examination or by history by extensive external lesions. Volunteers with a history of recurrent genital herpes disease characterized by limited external lesions are eligible to participate in the study.
* Positive tests for hepatitis C antibody, hepatitis B surface antigen, or HIV-1 antibody
* Any prior receipt of any vaccine (experimental or otherwise) for treatment or prophylaxis of genital warts or other papillomavirus related condition. Any treatment of genital warts or other papillomavirus related condition within 6 months of randomization (local therapy for common skin and/or plantar warts is allowed)
* Previous administration of any components of the investigational vaccine
* Receipt of any experimental vaccine within 90 days prior to entry into this study
* Receipt of any experimental drug therapy within 30 days or five half-lives of the experimental drug (if the half-life is known), whichever is longer

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2000-10; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Solicited adverse event rates (including injection site and systemic reactions) | For 7 days after each injection
Solicited adverse event rates | For 30 days after each injection
Serious adverse event rates | From first injection through 6 months after last injection
Laboratory assessments (Chemistry and Hematology parameters) | Study Days 0, 30 and 210
Vital signs (temperature, blood pressure, pulse rate, respiratory rate) | At the time of each injection and 30 minutes after each injection
Serum ELISA titers against HPV-16 and HPV-18 | 30 days after the third injection

SECONDARY OUTCOMES:
Serum ELISA titers against HPV-16 and HPV-18 | Study Days 0, 7, 30, 60, 180, 210, and 360, and at 18, 24, 36, and 48 months
Neutralization titers against HPV-16 and HPV-18 | Study Days 0, 60, 210 and 360
Inhibitory ELISAs | Study Days 0, 60, 210, and 360, and at 18, 24, 36, and 48 months
Lymphoproliferative, IL-5, and IFN-γ assays | Study Days 0, 60, 210, and 360, and at 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Descamps D, Hardt K, Spiessens B, Izurieta P, Verstraeten T, Breuer T, Dubin G. Safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine for cervical cancer prevention: a pooled analysis of 11 clinical trials. Hum Vaccin. 2009 May;5(5):332-40. doi: 10.4161/hv.5.5.7211. Epub 2009 May 20. PMID 19221517
- [Background] Giannini SL, Hanon E, Moris P, Van Mechelen M, Morel S, Dessy F, Fourneau MA, Colau B, Suzich J, Losonksy G, Martin MT, Dubin G, Wettendorff MA. Enhanced humoral and memory B cellular immunity using HPV16/18 L1 VLP vaccine formulated with the MPL/aluminium salt combination (AS04) compared to aluminium salt only. Vaccine. 2006 Aug 14;24(33-34):5937-49. doi: 10.1016/j.vaccine.2006.06.005. Epub 2006 Jun 19. PMID 16828940
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 580299/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 580299/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 580299/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 580299/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 580299/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 580299/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 580299/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register